CLINICAL TRIAL: NCT06883032
Title: Validation of the QuickSee Plus Device
Brief Title: Investigation of the Accuracy of an Automated Refractor to Provide Well-tolerated Eyeglass Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PlenOptika, Inc. (Industry)
Collaborators: New England College of Optometry (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Shivang R. Dave, PhD, CEO & co-founder, PlenOptika, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QuickSee Plus Trial; 2R44EY025452-04 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Refractive Errors
Keywords: refractive errors; eyeglasses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AR Eyeglasses, then SR Eyeglasses (Other): Automated Refraction (AR) Eyeglasses, then Subjective Refraction (SR) Eyeglasses
  Interventions: Other: AR Eyeglasses first, SR Eyeglasses second
- SR Eyeglasses, then AR Eyeglasses (Other): Subjective Refraction (SR) Eyeglasses, then Automated Refraction (AR) Eyeglasses
  Interventions: Other: SR Eyeglasses first, AR Eyeglasses second

INTERVENTIONS:
Other: AR Eyeglasses first, SR Eyeglasses second — First Eyeglasses based on Automated Refraction, Second Eyeglasses based on Subjective Refraction
  Arms: AR Eyeglasses, then SR Eyeglasses
Other: SR Eyeglasses first, AR Eyeglasses second — First Eyeglasses based on Subjective Refraction, Second Eyeglasses based on Automated Refraction
  Arms: SR Eyeglasses, then AR Eyeglasses

SUMMARY:
At the New England College of Optometry in Boston, MA, subjects ages 18-65 who have received or are receiving treatment for refractive error who choose to enroll in the study will be evaluated using subjective refraction and automated refraction, by way of the QuickSee Plus refractor. Subjects will then be randomized into one of two treatment plans: receive glasses from automated refraction first then subjective refraction second, and vice versa. After one week of wearing the first pair of glasses, patient preferences are assessed, and glasses are switched. After a week of wearing the second pair of glasses from the alternate measurement method, patient preferences are again assessed. Patients may then decide which pair patient like best. This is a triple blind, case-crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* who have had an eye exam at the NECO Center for Eye Care of Commonwealth or Roslindale
* who are aged between 18 years and 65 years

Exclusion Criteria:

* whose refractive error is outside of the detection range of the QuickSee Free Pro and QuickSee Plus devices: -13 D to +10 D (S) and -8 D to + 8 D (C)
* who are unable to provide consent
* who have undergone any eye surgery
* who have a history of ocular disease
* who are taking systemic drugs
* who wear more than one pair of single vision eyeglasses for distance
* who more than occasionally wear soft contact lenses
* who are unable and unwilling to wear the eyeglasses provided by the study for the required duration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Patient Preference | 2 weeks
  Patients are asked the question "Which eyeglasses did you prefer?". Patient response is then recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- New England College of Optometry (NECO) Center for Eye Care of Commonwealth, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: March 2025 - May 2025
Access Criteria: PlenOptika, New England College of Optometry, Data Safety Monitoring Board

REFERENCES:
- [Background] Joseph S, Varadaraj V, Dave SR, Lage E, Lim D, Aziz K, Dudgeon S, Ravilla TD, Friedman DS. Investigation of the Accuracy of a Low-Cost, Portable Autorefractor to Provide Well-Tolerated Eyeglass Prescriptions: A Randomized Crossover Trial. Ophthalmology. 2021 Dec;128(12):1672-1680. doi: 10.1016/j.ophtha.2021.05.030. Epub 2021 Jun 7. PMID 34111444